CLINICAL TRIAL: NCT04169269
Title: Patient Adherence to Venous Thromboembolism Prophylaxis in Orthopaedic Trauma Patients: A Randomized, Controlled Trial Comparing Subcutaneous Enoxaparin & Oral Rivaroxaban
Brief Title: Deep Vein Thrombosis Prophylaxis Adherence: Enoxaparin vs Rivaroxaban
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Florida Orthopaedic Institute (Network)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Principal Investigator, Barbara Steverson, Director of Research, Orthopaedic Trauma Service, Florida Orthopaedic Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20192684
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Deep Vein Thrombosis; Venous Thromboembolism
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism | interventions — Enoxaparin; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two medications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enoxaparin (Active Comparator): enoxaparin injectable, 40 milligram subcutaneous injection daily for 20 days
  Interventions: Drug: Enoxaparin 40 milligram/0.4 milliliter Injectable Syringe 0.4 milliliters
- Rivaroxaban (Active Comparator): rivaroxaban oral 10 milligram tablet daily for 20 days
  Interventions: Drug: Rivaroxaban 10 milligram Oral Tablet

INTERVENTIONS:
Drug: Enoxaparin 40 milligram/0.4 milliliter Injectable Syringe 0.4 milliliters — anticoagulant, subcutaneous injection
  Other Names: Lovenox
  Arms: Enoxaparin
Drug: Rivaroxaban 10 milligram Oral Tablet — anticoagulant, oral
  Other Names: Xarelto
  Arms: Rivaroxaban

SUMMARY:
The objective of this study is to compare oral rivaroxaban with injectable enoxaparin in orthopaedic trauma patients to determine if orally administered rivaroxaban once daily carries greater compliance and overall satisfaction than enoxaparin self-administered by subcutaneous injection once daily.

DETAILED DESCRIPTION:
This study is a randomized, controlled trial of orthopaedic trauma patients presenting to a single academic level one trauma center that require an extended course of venous thromboembolism event chemoprophylaxis. The goal is to compare oral rivaroxaban with our standard-of-care, injectable enoxaparin in orthopaedic trauma patients to determine if orally administered rivaroxaban once daily carries greater compliance and overall satisfaction than enoxaparin self-administered by subcutaneous injection once daily.

All patients included in the study would be treated with the standard enoxaparin 40 milligram injection while an inpatient. Upon hospital discharge, those requiring extended venous thromboembolism event chemoprophylaxis will be randomized to receive 20 days of either self-injected enoxaparin 40 milligrams or oral rivaroxaban,10 milligrams, a non-vitamin K oral anticoagulant. Both groups will then receive our current standard of care, aspirin 81 milligrams once daily for the remaining 3 weeks, for a total of 6 weeks of venous thromboembolism event chemoprophylaxis. Routine postoperative care will be provided by the treating surgeon.

ELIGIBILITY:
Inclusion Criteria:

* • Orthopaedic trauma patients deemed by the attending, treating surgeon to require an extended duration of venous thromboembolism chemoprophylaxis beyond that provided as an inpatient.

  * Patients being discharged directly to home.

Exclusion Criteria:

* • Patients being discharged to a rehabilitation center or a skilled nursing facility.

  * A contraindication to anticoagulation such as traumatic or other hemorrhage, as determined by the treating surgeon and/or consulting services.
  * Ongoing venous thromboembolism treatment or extended prophylaxis (i.e. past history of multiple deep vein thrombosis/pulmonary embolism) for current or recent deep vein thrombosis, pulmonary embolism or other coagulopathic disorder
  * Chronic anticoagulation for atrial fibrillation or other medical disorder requiring chronic anticoagulation therapy.
  * Perceived low-risk patients requiring only aspirin or no pharmacological venous thromboembolism prophylaxis.
  * Pregnant, prisoner, under 18 years old, or do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
adherence to medication regimen | 2 weeks
  measured with Morisky Medication Adherence Scale instrument; Score range is 0-8, 0 = low adherence to medication regimen, 8 = jigh adherence to medication regimen
adherence to medication regimen | 6 weeks
  measured with Morisky Medication Adherence Scale instrument; Score range is 0-8, 0 = low adherence to medication regimen, 8 = jigh adherence to medication regimen
patient satisfaction with treatment regimen | 2 weeks
  measured with Treatment Satisfaction Questionnaire for Medication (TSQM-9) instrument. TSQM-9 scores have a range of 0 to 100, with higher scores indicating higher satisfaction.
patient satisfaction with treatment regimen | 6 weeks
  measured with Treatment Satisfaction Questionnaire for Medication (TSQM-9) instrument. TSQM-9 scores have a range of 0 to 100, with higher scores indicating higher satisfaction.

SECONDARY OUTCOMES:
Number of participants with a bleeding event | 2 weeks
  measured through record review and participant reporting
Number of participants with a bleeding event | 6 weeks
  measured through record review and participant reporting
Number of participants with a bleeding event | 3 months
  measured through record review and participant reporting
Number of participants with a clotting event | 2 weeks
  measured through record review and participant reporting
Number of participants with a clotting event | 6 weeks
  measured through record review and participant reporting
Number of participants with a clotting event | 3 months weeks
  measured through record review and participant reporting
treatment cost | 3 months
  cost in U.S. dollars for 20 days of treatment drug

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Mir, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (1):
- Florida Orthopaedic Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] John MP 2nd, Streufert BD, Downes K, Chase CB, Mir HR. A Prospective Randomized Controlled Trial Comparing Enoxaparin & Rivaroxaban for Venous Thromboembolism Prophylaxis in Orthopaedic Trauma. J Orthop Trauma. 2022 Dec 1;36(12):615-622. doi: 10.1097/BOT.0000000000002454. PMID 36399673